CLINICAL TRIAL: NCT02571296
Title: The Value of Oral Micronized Progesterone in the Prevention of Spontaneous Preterm Birth
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ghamra Military Hospital (Other)
Collaborators: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Adel Abdel-Aziz, Registrar of OB/GYN, Ghamra Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 310
Record Dates: First submitted 2015-10-01; First posted 2015-10-08 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Preterm Birth
Keywords: Preterm Birth; Oral Micronized Progesterone
MeSH Terms: conditions — Premature Birth | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Active Comparator): subjects will recieve twice daily tablets of 100 mg of oral Micronized Progesterone from (14-18 weeks) until 36 weeks or delivery.
  Subjects: 106 cases Name: Oral micron ized progesterone Form: oral tablets Dosage: one tablet Frequency: every 12 hours Duration: 14-36 weeks gestational age.
  Interventions: Drug: micronized progesterone
- Group B (Placebo Comparator): subjects will receive placebo twice daily from (14-18 weeks) until 36 weeks or delivery.
  Subjects: 106 cases Name: placebo Form: oral tablets Dosage: one tablet Frequency: every 12 hours Duration: 14-36 weeks gestational age.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: micronized progesterone — Oral
  Other Names: Uterocare
  Arms: group A
Drug: Placebo — Oral
  Arms: Group B

SUMMARY:
This is a randomized, double-blind, placebo-controlled study.

DETAILED DESCRIPTION:
Intervention:

The study subjects will be randomized to receive twice daily tablets of either 100 mg of OMP (Uterocare®, October Pharma , Sixth of October city, Egypt) or placebo from enrollment (14-18 weeks) until 36 weeks or delivery, whichever occurs first. The patients and medical staff will be blinded to the study medication allocation.

Method of Randomization:

All patients who are fit for admission into the study will pull one of the numbered sealed identical black bags containing either the active medicine (=25%), the placebo (with the aim of admission into data collection, =25%), or a placebo together with a short note explaining that they will not be admitted to the study (=50%) and that they can give back their bag to the head nurse.

The code for the 424 (106x4) bag numbers is a confidential computer generated random number list (generated using MedCalc© Software bvba, Ostend, Belgium). It will be left, in a sealed envelope, with the head nurse of the antenatal clinic, till the end of data collection.ruptured membranes.

5. Obstetric ultrasound for gestational age, amniotic fluid volume, fetal weight, placental position, fetal anomalies.

6. Transvaginal ultrasound is not always available for cervical length assessment in ASUMH, so it will not be a necessary step in patients assessment but will be done whenever available.

Follow up:

Patients will be followed up regularly, at twice monthly intervals, in the antenatal clinic of Ain Shams University Maternity Hospital until delivery. They will be instructed to return to the hospital when recurrence of symptoms of preterm labor, rupture of membranes, or vaginal bleeding. There will be telephone call follow ups routinely to ensure adherence to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancies.
2. Gestational age, on admission, is between 14 and 18 weeks.
3. Past history of at least one idiopathic preterm birth.

Exclusion Criteria:

1. Established preterm labor (cervical dilatation ≥ 4 cm).
2. Persistent uterine contractions.
3. Women with medical or surgical complications indicating delivery or termination of pregnancy.
4. Presence of fetal anomalies incompatible with life.
5. Premature rupture of membranes.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 212 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The rate (incidence) of preterm delivery (gestational age <37 weeks). | up to 37weeks.
  Patients will be followed up regularly, at twice monthly intervals, in the antenatal clinic of Ain Shams University Maternity Hospital until delivery. They will be instructed to return to the hospital when recurrence of symptoms of preterm labor, rupture of membranes, or vaginal bleeding. There will be telephone call follow up routinely to ensure adherence to the study protocol.

SECONDARY OUTCOMES:
The incidence of rupture of the amniotic membranes. | up to 37weeks.
  Patients will be followed up regularly, at twice monthly intervals, in the antenatal clinic of Ain Shams University Maternity Hospital until delivery. They will be instructed to return to the hospital when recurrence of symptoms of preterm labor, rupture of membranes, or vaginal bleeding. There will be telephone call follow up routinely to ensure adherence to the study protocol.
The neonatal birth weight | up to 37 weeks.
  Patients will be followed up regularly, at twice monthly intervals, in the antenatal clinic of Ain Shams University Maternity Hospital until delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdel-Aziz, Principal Investigator — Ain Shams Maternity Hospital
Locations (1):
- Ahmed Adel Abdel-Aziz, Cairo, Egypt